CLINICAL TRIAL: NCT03100552
Title: Prediction of Dysplasia Within Sessile Serrated Polyps Using Endoscopic Imaging; a Prospective Observational Study
Acronym: SERRESH
Status: Completed | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Clinical Professor of Medicine, Western Sydney Local Health District
Other Study IDs: 4075
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Sessile Serrated Adenoma
Keywords: Colonoscopy; Endoscopic resection; Sessile serrated adenoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Patients referred to a tertiary endoscopic resection practice found to have an SSP >= 8mm. Endoscopic imaging applied to the sessile serrated polyp (SSP) to determine the presence or absence of dysplasia.
  Interventions: Diagnostic Test: Endoscopic imaging

INTERVENTIONS:
Diagnostic Test: Endoscopic imaging — Analysis of the presence of dysplasia within sessile serrated polyps (SSP) using endoscopic imaging (high definition white light +- narrow band imaging)

SUMMARY:
Study of endoscopic imaging in the detection of dysplasia within serrated colonic lesions >= 8mm in size

DETAILED DESCRIPTION:
Observational study Structured endoscopic imaging protocol devised Applied prospectively to sequential SSP >= 8mm detected in a tertiary endoscopic resection cohort Review of specimens by blinded specialist pathologists Review of incongruent cases by endoscopists and pathologists

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to a tertiary endoscopic resection practice with any sessile serrated polyp (SSP) >= 8mm

Exclusion Criteria:

* Patients referred to a tertiary endoscopic resection practice without sessile serrated polyps (SSP)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to a tertiary endoscopic resection practice with any SSP >= 8mm
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Dysplasia | at the initial procedure when the sessile serrated polyp (SSP) is analysed by the endoscopist compared with when the SSP is analysed at histopathology less than one week later. no ongoing determination
  Presence of dysplasia within sessile serrated polyps (SSP) using endoscopic imaging and congruence with histopathology

SECONDARY OUTCOMES:
Sessile serrated polyp | at the initial procedure compared with histopathology within 1 week. no ongoing determination
  Determination of a specific polyp as an sessile serrated polyp (SSP)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, MBBS, FRACP, Principal Investigator — WSLHD
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tate DJ, Jayanna M, Awadie H, Desomer L, Lee R, Heitman SJ, Sidhu M, Goodrick K, Burgess NG, Mahajan H, McLeod D, Bourke MJ. A standardized imaging protocol for the endoscopic prediction of dysplasia within sessile serrated polyps (with video). Gastrointest Endosc. 2018 Jan;87(1):222-231.e2. doi: 10.1016/j.gie.2017.06.031. Epub 2017 Jul 13. PMID 28713060